CLINICAL TRIAL: NCT01589692
Title: A Clinical Trial for the Surgical Treatment of Elderly Distal Radius Fractures. The Wrist and Radius Injury Surgical Trial (WRIST)
Brief Title: A Clinical Trial for the Surgical Treatment of Elderly Distal Radius Fractures
Acronym: WRIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dr. Kevin C. Chung, Charles B. G. de Nancrede Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR062066-01A1 (NIH); R01AR062066-01A1 (NIH)
Record Dates: First submitted 2012-04-25; First posted 2012-05-02 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Distal Radius Fracture
Keywords: WRIST; Distal Radius Fracture; DRF; elderly; internal fixation; VLPS; External Fixation; Multi center randomized trial
MeSH Terms: conditions — Wrist Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal; External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Internal Fixation (Experimental): Open Reduction and Internal Fixation: Internal fixation with a volar locking plating system
  Interventions: Procedure: Open Reduction and Internal Fixation
- External Fixation (Experimental): External Fixation with a bridging external fixator. Can be done with or without percutaneous pinning.
  Interventions: Procedure: External Fixation
- Pinning (Experimental): Percutaneous pinning with any number of Kirschner wires
  Interventions: Procedure: Percutaneous Pinning
- No Surgery (Active Comparator): Closed Reduction and casting: Closed reduction and immobilization with a cast and/or splint
  Interventions: Procedure: Closed Reduction and casting

INTERVENTIONS:
Procedure: Open Reduction and Internal Fixation — Internal fixation with a volar locking plating system
  Arms: Internal Fixation
Procedure: External Fixation — External Fixation with a bridging external fixator. Can be done with or without percutaneous pinning.
  Arms: External Fixation
Procedure: Percutaneous Pinning — Pinning with any number of Kirschner wires
  Arms: Pinning
Procedure: Closed Reduction and casting — Closed reduction and immobilization with a cast and/or splint
  Arms: No Surgery

SUMMARY:
In the United States, over 300,000 individuals over age 65 suffer from distal radius fractures (DRFs) each year. Despite the frequency of this injury and over 200 years of experience treating DRFs, management of elderly DRFs is still controversial. Close reduction and casting is a nonsurgical technique that is frequently used, but osteoporotic fractures, common in the elderly, often collapse and displace. The three currently applied surgical techniques are close reduction and percutaneous pinning, external fixation with or without percutaneous pinning, and internal fixation with volar locking plating. Preliminary evidence indicates that locking plate fixation can permit elderly patients to move their hands and wrists much sooner in order to return to self-care activities more quickly. Although these outcomes are promising, there is no randomized controlled clinical trial to demonstrate that the more invasive, and perhaps more costly, plating technique is superior to the other simpler approaches.

The specific aim of this 24-center randomized controlled trial is to compare outcomes of these three surgical techniques in treating unstable DRFs in the elderly. The secondary aim is to follow a cohort of elderly patients who choose not to have surgery to evaluate outcomes following treatment by close reduction and casting alone. This clinical trial is the most ambitious study in hand surgery by assembling most of the leading centers in North America to collect evidence-based data to guide future treatment of this prevalent injury in the growing elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an unstable DRF for which surgical fixation is indicated

  o AO type A2, A3, C1, C2
* At least one of the following radiographic criteria indicating fracture instability

  * Dorsal angulation of greater than 10°
  * Radial inclination angle of less than 15°
  * Radial shortening of greater than 3mm
* Patients with the ability to read and understand English (to complete study questionnaires)
* Community-dwelling patients
* Patients 60 years of age or older

Exclusion Criteria:

* Patients who have suffered open DRFs
* Patients with bilateral DRFs
* Patients with associated upper extremity fractures or ligament injuries (including ulnar styloid fracture, TFCC and wrist ligament injuries) requiring repair at the time of DRF fixation
* Multi-trauma patients
* Patients with prior DRF on the same wrist
* Patients with comorbid conditions prohibiting surgery
* Patients with neurologic disorders that affect hand, wrist or arm sensation or movement
* Patients who have a history of dementia, Alzheimer's Disease or other serious psychiatric disorders
* Patients with current substance abuse
* Patients who do not agree to be randomized
* Patients who have DRFs that are not equally suited for each procedure (i.e. severely comminuted fractures)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2012-04-10 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Michigan Hand Outcomes Questionnaire score | 12months
  upper-extremity questionnaire

SECONDARY OUTCOMES:
Change in Rapid Assessment of Physical Activity score | pre-injury and 24months
  questionnaire
SF-36 score | 12months
  QOL questionnaire
complications | 12months
  Complication Checklist for Distal Radius Fracture
Hand function | 12months
  grip strength, lateral pinch strength, wrist motion

OTHER OUTCOMES:
Participant Demographics | baseline
  Participant age, income, education level, race/ethnicity
Comorbidities | baseline
  Self-Administered Comorbidity Checklist
Therapy compliance | 12months
  count of therapy sessions and description of therapy type

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Chung, MD, MS, Principal Investigator — University of Michigan
Locations (24):
- United States (20):
  - University of Connecticut, Farmington, Connecticut
  - Norton Healthcare, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - HealthPartners Institute for Education and Research, Saint Paul, Minnesota
  - North Shore - Long Island Jewish Health System, Great Neck, New York
  - University of Rochester, Rochester, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Kettering Health Network, Centerville, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
- Canada (3):
  - Fraser Health Authority, New Westminster, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - University of Western Ontario, London, Ontario
- National University of Singapore, Singapore, Singapore

REFERENCES:
- [Background] Chung KC, Song JW; WRIST Study Group. A guide to organizing a multicenter clinical trial. Plast Reconstr Surg. 2010 Aug;126(2):515-523. doi: 10.1097/PRS.0b013e3181df64fa. PMID 20375760
- [Background] Wrist and Radius Injury Surgical Trial (WRIST) Study Group. Reflections 1 year into the 21-Center National Institutes of Health--funded WRIST study: a primer on conducting a multicenter clinical trial. J Hand Surg Am. 2013 Jun;38(6):1194-201. doi: 10.1016/j.jhsa.2013.02.027. Epub 2013 Apr 20. PMID 23608306
- [Derived] Jayaram M, Wu H, Yoon AP, Kane RL, Wang L, Chung KC. Comparison of Distal Radius Fracture Outcomes in Older Adults Stratified by Chronologic vs Physiologic Age Managed With Casting vs Surgery. JAMA Netw Open. 2023 Feb 1;6(2):e2255786. doi: 10.1001/jamanetworkopen.2022.55786. PMID 36780156
- [Derived] Yoon AP, Wang Y, Wang L, Chung KC; and the WRIST Group. What Are the Tradeoffs in Outcomes after Casting Versus Surgery for Closed Extraarticular Distal Radius Fractures in Older Patients? A Statistical Learning Model. Clin Orthop Relat Res. 2021 Dec 1;479(12):2691-2700. doi: 10.1097/CORR.0000000000001865. PMID 34142664
- [Derived] Chung KC, Kim HM, Malay S, Shauver MJ; WRIST Group. Comparison of 24-Month Outcomes After Treatment for Distal Radius Fracture: The WRIST Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2112710. doi: 10.1001/jamanetworkopen.2021.12710. PMID 34137830
- [Derived] Yoon AP, Wang C, Speth KA, Wang L, Chung KC; WRIST Group. Modifiable Factors Associated With Chronic Pain 1 Year After Operative Management of Distal Radius Fractures: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2028929. doi: 10.1001/jamanetworkopen.2020.28929. PMID 33337492
- [Derived] Hooper RC, Zhou N, Wang L, Shauver MJ, Chung KC; WRIST Group. Pre-injury activity predicts outcomes following distal radius fractures in patients age 60 and older. PLoS One. 2020 May 20;15(5):e0232684. doi: 10.1371/journal.pone.0232684. eCollection 2020. PMID 32433648
- [Derived] Chung KC, Cho HE, Kim Y, Kim HM, Shauver MJ; WRIST Group. Assessment of Anatomic Restoration of Distal Radius Fractures Among Older Adults: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Jan 3;3(1):e1919433. doi: 10.1001/jamanetworkopen.2019.19433. PMID 31951273
- [Derived] Chung KC, Malay S, Shauver MJ, Kim HM; WRIST Group. Assessment of Distal Radius Fracture Complications Among Adults 60 Years or Older: A Secondary Analysis of the WRIST Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e187053. doi: 10.1001/jamanetworkopen.2018.7053. PMID 30657531
- [Derived] Nasser JS, Huetteman HE, Shauver MJ, Chung KC. Older Patient Preferences for Internal Fixation after a Distal Radius Fracture: A Qualitative Study from the Wrist and Radius Injury Surgical Trial. Plast Reconstr Surg. 2018 Jul;142(1):34e-41e. doi: 10.1097/PRS.0000000000004454. PMID 29952895